CLINICAL TRIAL: NCT07228390
Title: A PHASE 2, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, 16-WEEK STUDY EVALUATING THE SAFETY AND EFFICACY OF RITLECITINIB (PF-06651600) IN ADULTS WITH MODERATE TO SEVERE HIDRADENITIS SUPPURATIVA
Brief Title: A 16-Week Study to Learn About the Study Medicine Called Ritlecitinib in Adults With Long Lasting Painful Red Skin Lumps, Known by the Medical Term, Hidradenitis Suppurativa, or HS.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7981119; 2025-522705-37-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-10-31; First posted 2025-11-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Ritlecitinib
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Intervention (Experimental): Participants will receive one oral dose once daily (QD), starting with a loading dose of ritlecitinib for 8 weeks, followed by maintenance for 8 weeks.
  Interventions: Drug: Ritlecitinib
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritlecitinib — Participants will receive one oral dose once daily (QD), starting with a loading dose of ritlecitinib for 8 weeks, followed by maintenance for 8 weeks.
  Other Names: Investigational Product
  Arms: Study Intervention
Drug: Placebo — Participant will receive matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called Ritlecitinib) for the possible treatment of hidradenitis suppurativa (HS). HS is a disease causing long lasting painful red skin lumps.

This study is seeking participants who:

* have moderate or severe HS
* have previously received antibiotics for HS that did not help, or could not tolerate antibiotics Participants will be randomly (like a flip of coin) assigned to receive either the study medicine or a placebo (a pill that looks like the study medicine but does not contain any medicine). The study medicine or placebo will be taken by mouth once daily at home. For the first part of the study, participants will receive a loading (starting) dose. For the next part of the study, participants will receive a maintenance (ongoing) dose.

Participants will take part in the study for about 24 weeks (about 6 months). There will be about 10 study clinic visits: a screening visit, Day 1, and then every 1, 2, or 4 weeks until week 16. At each visit, participants will report on their health and have tests such as physical exams, blood and urine tests, vital signs, chest X-rays, ECGs, hearing tests, and questionnaires. Participants will record when they take the study medicine and their HS symptoms every day in an eDiary on a mobile phone.

The experiences of participants receiving the study medicine will be compared to those receiving placebo to help see if the study medicine is safe and effective.

ELIGIBILITY:
Key Eligibility Criteria:

Inclusion Criteria:

1. Male or female participants ≥18 to ≤75 years of age.
2. Participants with a diagnosis (based on clinical history and physical examination) of moderate to severe HS for at least 6 months prior to Screening Visit and inadequate response to at least 4-week (28 days) treatment with oral antibiotics for the treatment of HS.

Exclusion Criteria:

1. Presence of ≥20 draining fistulae at Screening or BL visit
2. Evidence of other active skin disease or condition at screening
3. Have a known immunodeficiency disorder
4. Having a history of systemic infection requiring hospitalization or parenteral therapy, including history of infection with Mycobacterium TB
5. Specific Viral Infection History (incl. history of herpes zoster, HBV or HCV Infection
6. Current or recent history of clinically significant severe, progressive, or uncontrolled other medical conditions
7. Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-03-05 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of responders based on Hidradenitis Suppurativa Clinical Response achieving at least 50% reduction from baseline (Hidradenitis Suppurativa Clinical Response HiSCR50) in patients with HS treated with ritlecitinib versus placebo. | Week 16
  The difference in proportion of responders based on HiSCR50 response at Week 16 in patients with HS treated with ritlecitinib versus placebo.

SECONDARY OUTCOMES:
Proportion of participants achieving HiSCR50 response | at Weeks 1, 2, 4, 6, 8 and Week 12.
  The difference in proportion of responders based on HiSCR50 response at Weeks 1, 2, 4, 6, 8 and 12 in patients with HS treated with ritlecitinib versus placebo
Proportion of participants achieving HiSCR75 response | at Weeks 1, 2, 4, 6, 8, 12 and Week 16.
  The difference in proportion of responders based on HISCR75 response at Weeks 1, 2, 4, 6, 8, 12 and 16 in patients with HS treated with ritlecitinib versus placebo
Proportion of participants achieving HiSCR90 response | at Weeks 1, 2, 4, 6, 8, 12 and Week 16
  The difference in proportion of responders based on HiSCR90 response at Weeks 1, 2, 4, 6, 8, 12 and 16 in patients with HS treated with ritlecitinib versus placebo
Response based on a on total abscess and inflammatory nodule count (AN Count) of 0 or 1 | Week 16
  The difference in proportion of responders based on a total AN count of 0 or 1 at Week 16 in patients with HS treated with ritlecitinib and placebo
Response based on a total AN count of 0, 1, or 2 | At week 16
  The difference in proportion of responders based on a total AN count of 0, 1 or 2 at Week 16 in patients with HS treated with ritlecitinib and placebo.
Percent change from Baseline(CFB) in total AN count | Weeks 1, 2, 4, 6, 8, 12 and 16.
  The difference in mean percent CFB in total AN count at Weeks 1, 2, 4, 6, 8, 12 and 16 in patients with HS treated with ritlecitinib and placebo
Absolute score in Hidradenitis Suppurativa Investigator Global Assessment (HS-IGA) | at Weeks 1, 2, 4, 6, 8, 12 and 16
  The difference in mean absolute score in HS-IGA at Weeks 1, 2, 4, 6, 8, 12 and 16 in patients with HS treated with ritlecitinib and placebo
CFB in Hidradenitis Suppurativa Investigator Global Assessment (HS-IGA) | at Weeks 1, 2, 4, 6, 8, 12 and 16
  Mean CFB in HS-IGA at Weeks 1, 2, 4, 6, 8, 12 and 16 in patients with HS treated with ritlecitinib and placebo
Proportion of participants achieving a HS-IGA=0 or 1 | Weeks 1, 2, 4, 6, 8, 12 and 16
  The difference in proportion of responders based on HS-IGA=0 or 1 at Weeks 1, 2, 4, 6, 8, 12 and 16 in patients with HS treated with ritlecitinib and placebo
Participants who experience an HS flare, defined as at least a 25% increase in total AN count with a minimum increase of 2 relative to Baseline | Weeks 4, 8, 12 and 16.
  The difference in proportion of HS flare at Weeks 4, 8, 12 and 16 in patients with HS treated with ritlecitinib and placebo
CFB in Hidradenitis Suppurativa Symptom Daily Diary (HSSDD) | Weeks 1, 2, 4, 6, 8, 12 and 16
Skin pain NRS30 (numeric rating scale) response, at worst and on average, respectively among participants with baseline skin pain NRS ≥3 | Weeks 1, 2, 4, 6, 8, 12, and 16
Percent CFB in skin pain NRS, at worst and on average, respectively, in participants with baseline skin pain NRS ≥3 | Weeks 1, 2, 4, 6, 8, 12, and 16
CFB in skin pain NRS, at worst and on average, respectively | at Weeks 1, 2, 4, 6, 8, 12, and 16
Skin pain NRS50 response, at worst and on average, respectively among participants with baseline skin pain NRS ≥3. | at Weeks 1, 2, 4, 6, 8, 12, and 16
Skin pain NRS70 response, at worst and on average, respectively among participants with baseline skin pain NRS ≥3 | at Weeks 1, 2, 4, 6, 8, 12, and 16,
Incidence of treatment emergent adverse events (TEAE), adverse events (AE) and serious adverse events (SAE) leading to discontinuation | up to 24 Weeks
Incidence of clinically significant laboratory abnormalities over time | up to 24 Weeks
Absolute score and CFB in Hidradenitis Suppurativa Quality of Life (HiSQOL) | at Weeks 1, 2, 4, 6, 8, 12 and 16.
Absolute score and % CFB in International Hidradenitis Suppurativa Severity Score System (IHS4) | Weeks 1, 2, 4, 6, 8, 12 and 16.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Northridge Clinical Trials, Northridge, California
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Revival Research Institute, LLC, Troy, Michigan
  - ClinOhio Research Services, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981119